CLINICAL TRIAL: NCT05620784
Title: Loop Diuretics During Morcellation to Improve Same-day Discharge Rates After Holmium Laser Enucleation of the Prostate (HoLEP)
Brief Title: Intra-operative Loop Diuretics to Improve Same-day Discharge Rates After HoLEP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Director of The Division of Endourology & Stone Disease, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00217795
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: BPH With Urinary Obstruction; BPH; Hematuria; Same Day Discharge
MeSH Terms: conditions — Hematuria | interventions — Furosemide; Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1
Who Masked: Participant, Care Provider
Masking Description: Only the clinical investigator and anesthesiologist/nurse anesthetist will be aware of treatment allocation. The care providers (surgeon, fellow, resident, and nursing team) and patient will be blinded to the treatment allocation. The outcomes assessor will be unblinded at the time of statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Loop Diuretic (Furosemide) (Experimental): This group of patients will receive 20mg of IV furosemide during the morcellation phase of their HoLEP.
  Interventions: Drug: Furosemide
- Control (No Intervention): This group of patients will not receive 20mg of IV furosemide during the morcellation phase of their HoLEP.

INTERVENTIONS:
Drug: Furosemide — 20mg of IV furosemide injection during the morcellation phase of HoLEP
  Other Names: Lasix; Loop diuretic
  Arms: Loop Diuretic (Furosemide)

SUMMARY:
Holmium Laser Enucleation of the Prostate (HoLEP) is a size-independent treatment option for benign prostatic hypertrophy (BPH) as recommended by the American Urological Association (AUA) Guidelines. Loop diuretics (furosemide) have been given historically during the morcellation portion of HoLEP to promote urine production in the post-operative setting and to minimize the impact of fluid absorption during long periods of morcellation. The intra-operative use of 20mg IV furosemide in perioperative HoLEP pathways has been propagated with the dissemination of HoLEP across North America without evidence to support its routine administration. With increasing surgical efficiency from improvements in laser and morcellator technology, the role of intra-operative furosemide is unknown. This study is designed to assess if there is a significant difference in same day discharge rates after Holmium Laser Enucleation of the Prostate (HoLEP) with and without IV furosemide. .

DETAILED DESCRIPTION:
Holmium Laser Enucleation of the Prostate (HoLEP) is a size-independent treatment option for benign prostatic hypertrophy (BPH) as recommended by the American Urological Association (AUA) Guidelines. Loop diuretics (furosemide) have been given historically during the morcellation portion of HoLEP to promote urine production in the post-operative setting and to minimize the impact of fluid absorption during long periods of morcellation. The intra-operative use of 20mg IV furosemide in perioperative HoLEP pathways has been propagated with the dissemination of HoLEP across North America without evidence to support its routine administration.

This single-center randomized controlled trial is designed to assess if there is a significant difference in same day discharge rates after Holmium Laser Enucleation of the Prostate (HoLEP). We currently attempt to perform HoLEP as a same-day discharge (SDD) procedure, however one of the main limiting factors in SDD is hematuria. Loop diuretics (furosemide) have been administered at the time of morcellation as a part of our HoLEP pathway to increase post-operative urinary output and reduce clinically significant gross hematuria and clot-formation. The objective of our study will be to assess if SDD rates are non-inferior in those patients who do not receive furosemide diuretics versus those that do.

Patients will be randomized 1:1 to 20mg of IV lasix versus control. Patients and the surgeon/post-operative care team (fellow, residents, and nursing team) will be blinded to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 -89 undergoing HoLEP
* Willing to sign the Informed Consent Form
* Able to read, understand, and complete patient questionnaires.

Exclusion Criteria:

* Allergy or hypersensitivity to furosemide or other loop diuretic
* Anuric patients or patients with liver failure
* Patients having a concurrent ureteroscopy +/- laser lithotripsy, percutaneous nephrolithotomy, or non-urologic surgery at the time of their HoLEP
* Anticipated need for perineal urethrostomy at the time of HoLEP
* Patient not undergoing catheter removal and voiding trial at Northwestern Memorial Hospital

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Same-day discharge | 90-days
  Rate of successful same-day discharge after HoLEP
Same-day catheter removals | 90-days
  Rate of successful same-day catheter removals after HoLEP

SECONDARY OUTCOMES:
Adverse medical events (hematuria) | 90-days
  Rate of unplanned Emergency Department (ED) visits/clinic visits related to bleeding/admission/clot evacuation
Adverse medical events (fluid absorption) | 90-days
  Rate of transurethral resection (TUR) syndrome, vision changes, seizure, hyponatremia, electrolyte abnormality
Duration of post-operative hematuria | 90-days
  (days)
Difference in operative efficiency (enucleation, morcellation, and overall) | 90-days
  (minutes/gram)
Length of hospital stay | 90-days
  (hours)
Overall complications | 90-days
  Clavien-Dindo Classification

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Krambeck, MD, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parsons JK, Dahm P, Kohler TS, Lerner LB, Wilt TJ. Surgical Management of Lower Urinary Tract Symptoms Attributed to Benign Prostatic Hyperplasia: AUA Guideline Amendment 2020. J Urol. 2020 Oct;204(4):799-804. doi: 10.1097/JU.0000000000001298. Epub 2020 Jul 23. PMID 32698710
- [Background] Agarwal DK, Large T, Tong Y, Stoughton CL, Damler EM, Nottingham CU, Rivera ME, Krambeck AE. Same Day Discharge is a Successful Approach for the Majority of Patients Undergoing Holmium Laser Enucleation of the Prostate. Eur Urol Focus. 2022 Jan;8(1):228-234. doi: 10.1016/j.euf.2020.12.018. Epub 2021 Jan 4. PMID 33414073
- [Background] Kuo RL, Paterson RF, Kim SC, Siqueira TM Jr, Elhilali MM, Lingeman JE. Holmium Laser Enucleation of the Prostate (HoLEP): A Technical Update. World J Surg Oncol. 2003 Jun 6;1(1):6. doi: 10.1186/1477-7819-1-6. PMID 12818001
- [Background] Elzayat E, Habib E, Elhilali M. Holmium laser enucleation of the prostate in patients on anticoagulant therapy or with bleeding disorders. J Urol. 2006 Apr;175(4):1428-32. doi: 10.1016/S0022-5347(05)00645-2. PMID 16516015